CLINICAL TRIAL: NCT02833506
Title: A Phase I Clinical Trial of mTOR Inhibition With Sirolimus for Enhancing NY-ESO-1 Protein With MIS416 Vaccine Induced Anti-Tumor Immunity in Ovarian, Fallopian Tube and Primary Peritoneal Cancer
Brief Title: Sirolimus and Vaccine Therapy in Treating Patients With Stage II-IV Ovarian, Fallopian Tube, or Primary Peritoneal Cancer
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: production of adjuvant to be used with vaccine was discontinued by sponsor
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: I 277115; NCI-2016-00811 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 277115 (Other: RoswellPark); P30CA016056 (NIH); R01CA158318 (NIH)
Record Dates: First submitted 2016-07-08; First posted 2016-07-14 (Estimated); Last update posted 2018-05-01 (Actual); Status verified 2018-04

CONDITIONS: Recurrent Fallopian Tube Carcinoma; Recurrent Ovarian Carcinoma; Recurrent Primary Peritoneal Carcinoma; Stage IIA Fallopian Tube Cancer; Stage IIA Ovarian Cancer; Stage IIB Fallopian Tube Cancer; Stage IIB Ovarian Cancer; Stage IIC Fallopian Tube Cancer; Stage IIC Ovarian Cancer; Stage IIIA Fallopian Tube Cancer; Stage IIIA Ovarian Cancer; Stage IIIA Primary Peritoneal Cancer; Stage IIIB Fallopian Tube Cancer; Stage IIIB Ovarian Cancer; Stage IIIB Primary Peritoneal Cancer; Stage IIIC Fallopian Tube Cancer; Stage IIIC Ovarian Cancer; Stage IIIC Primary Peritoneal Cancer; Stage IV Fallopian Tube Cancer; Stage IV Ovarian Cancer; Stage IV Primary Peritoneal Cancer
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms | interventions — Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort I (NY-ESO-1 protein with MIS416) (Active Comparator): Patients receive NY-ESO-1 protein with MIS416 vaccine SC on days 1, 15, 29, 57, 85, and 113 in the absence of disease progression or toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Biological: Recombinant NY-ESO-1 Protein
- Cohort II (NY-ESO-1 protein with MIS416, sirolimus) (Experimental): Patients receive NY-ESO-1 protein with MIS416 vaccine as in Cohort I. Patients also receive sirolimus PO daily for 2 weeks followed by 2 weeks off starting on days 1, 29, 57, and 85.
  Interventions: Other: Laboratory Biomarker Analysis; Biological: Recombinant NY-ESO-1 Protein; Drug: Sirolimus

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Recombinant NY-ESO-1 Protein — Given recombinant NY-ESO-1 protein SC
Drug: Sirolimus — Given PO
  Other Names: AY 22989; RAPA; Rapamune; RAPAMYCIN; SILA 9268A; WY-090217
  Arms: Cohort II (NY-ESO-1 protein with MIS416, sirolimus)

SUMMARY:
This phase I clinical trial studies the side effects of sirolimus and NY-ESO-1 protein with MIS416 in treating patients stage II-IV ovarian, fallopian tube, or primary peritoneal cancer. Sirolimus may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Vaccine therapy, like Y-ESO-1 protein with MIS416, may strengthen the immune system to find and kill tumor cells. Biological therapies, such as sirolimus, use substances made from living organisms that may stimulate or suppress the immune system in different ways and stop tumor cells from growing. Giving sirolimus and vaccine therapy may work betting in treating patients with ovarian, fallopian tube or primary peritoneal cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Determine the safety and feasibility of NY-ESO-1 protein with MIS416 in combination with mammalian target of rapamycin (mTOR) inhibitor sirolimus.

SECONDARY OBJECTIVES:

I. To determine the effectiveness of these combinatorial therapies by assessing NY-ESO-1 specific cellular and humoral immunity: peripheral blood NY-ESO-1 specific cluster of differentiation (CD)8+ and CD4+ T-cells; peripheral blood NY-ESO-1 specific antibodies; peripheral blood frequency of CD4+ CD25+ forkhead box P3 (FOXP3)+ regulatory T-cells; explore time to disease progression.

OUTLINE:

COHORT I (C1): Patients receive NY-ESO-1 protein with MIS416 vaccine subcutaneously (SC) on days 1, 15, 29, 57, 85, and 113 in the absence of disease progression or toxicity.

COHORT II (C2): Patients receive NY-ESO-1 protein with MIS416 vaccine as in Cohort I. Patients also receive sirolimus orally (PO) daily for 2 weeks followed by 2 weeks off starting on days 1, 29, 57, and 85.

After completion of study treatment, patients are followed up at 30 days and then at 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Women with stages II-IV epithelial ovarian, fallopian tube, or primary peritoneal carcinoma who have completed standard therapy for primary or recurrent disease (i.e., patients who would normally be observed); eligible patients may have asymptomatic residual measurable disease on physical examination and/or computed tomography (CT) scan, and/or may have an elevated cancer antigen 125 (CA-125); or may be in complete clinical remission after treatment for primary or recurrent disease; these patients would normally enter a period of observation after standard management
* Any human leukocyte antigen (HLA) type (historic HLA typing is permitted)
* Tumor expression of NY-ESO-1 by immunohistochemistry (IHC) and/or real-time polymerase chain reaction (RTPCR)
* No history of previous severe allergic reactions to vaccines or unknown allergens
* Life expectancy > 6 months
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of =< 2
* Hematology and biochemistry laboratory results within the limits normally expected for the patient population, without evidence of major organ failure
* Absolute neutrophil count (ANC) >= 1,000/uL
* Platelets (PLT) >= 75,000/uL
* Hemoglobin (Hgb) >= 8 g/dL
* Total bilirubin =< 1.5 x upper limits of normal (ULN)
* Serum glutamic-oxaloacetic transaminase(SGOT)/aspartate aminotransferase (AST) or serum glutamate pyruvate transaminase(SGPT)/alanine aminotransferase (ALT) =< 3 x ULN
* Serum creatinine =< 2 x ULN
* Prothrombin time(PT)/international normalized ratio(INR) =< 1.5
* Electrocardiogram, showing no indications of cardiac problems like congestive heart failure, myocardial infarction, and cardiomyopathy
* Have been informed of other treatment options
* Ability to swallow and retain oral medication
* Participants of child-bearing potential must agree to use adequate contraceptive methods (e.g., hormonal or barrier method of birth control) prior to study entry; should a woman become pregnant or suspect she is pregnant while she is participating in this study, she should inform her treating physician immediately
* Participant or legal representative must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure
* Patients may have received previous NY-ESO-1 vaccine therapy

Exclusion Criteria:

* Metastatic disease to the central nervous system
* Other serious illnesses (e.g., serious infections requiring antibiotics, bleeding disorders)
* History of severe autoimmune disorders requiring use of steroids or other immunosuppressives
* Concomitant systemic treatment with corticosteroids, anti-histamine or non-steroidal antiinflammatory drugs for >2 weeks,, and other platelet inhibitory agents, strong inhibitors/inducers of cytochrome P450-3A4 (CYP450-3A4)
* Chemotherapy, radiation therapy, or immunotherapy within 4 weeks prior to first dosing of study drug (6 weeks for nitrosoureas); concomitant hormonal therapies for breast cancers are allowed
* Patients with a positive fecal occult blood test excluding hemorrhoids
* Clinically significant heart disease (New York Heart Association [NYHA] class III or IV) within six months
* Participation in any other clinical trial involving another investigational agent within 4 weeks prior to first dosing of study drug
* Known hepatitis B, hepatitis C, or human immunodeficiency virus (HIV)
* Mental impairment that may compromise the ability to give informed consent and comply with the requirements of the study
* Lack of availability of a patient for immunological and clinical follow-up assessment
* Known pulmonary hypertension
* Known hypersensitivity to sirolimus
* Evidence of current drug or alcohol abuse or psychiatric impairment, which in the Investigator's opinion will prevent completion of the protocol therapy or follow-up
* Pregnant or nursing female patients
* Unwilling or unable to follow protocol requirements
* Any condition which in the investigator's opinion deems the patient an unsuitable candidate to receive study drug (i.e., any significant medical illness or abnormal laboratory finding that would, in the investigator's judgment, increase the subject's risk by participating in this study)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-12-08 (Actual); Primary Completion 2018-08-15 (Estimated); Study Completion 2019-08-15 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events defined by National Cancer Institute Common Terminology Criteria for Adverse Events version 4.03 | Up to 30 days
  The toxicity rate for each adverse event will be estimated using a two-sided, 95%, exact binomial confidence interval (Clopper-Pearson).

SECONDARY OUTCOMES:
NY-ESO-1 specific CD4+ and CD8+ T-cells cellular immunity assessed in peripheral blood by enzyme-linked immunosorbent spot (ELISPOT) and intracellular cytokine staining (ICS) | Up to 12 months
  Assessed iin peripheral blood by enzyme-linked immunosorbent spot (ELISPOT) and intracellular cytokine staining (ICS)
NY-ESO-1 specific humoral immunity | Up to 12 months
  assessed in peripheral blood by ELISA
Time to disease progression as documented by Response Evaluation Criteria in Solid Tumors version 1.1 | Up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Kunle Odunsi, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States